CLINICAL TRIAL: NCT06729723
Title: A Multicenter, Randomized, Open-label, Parallel-group, Exploratory Clinical Trial to Evaluate the Effect of the Software as a Medical Device (SaMD) SAT-001 on the Changes in Choroidal Thickness in Pediatric Myopia Patients
Brief Title: Exploratory Study on the Effect of SAT-001 on Choroidal Thickness in Pediatric Myopia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: S-Alpha Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAT-001-KP-004
Record Dates: First submitted 2024-12-04; First posted 2024-12-11 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Myopia
Keywords: Myopia; Choroidal thickness; SaMD
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SAT-001 Treatment Group (Experimental): Using SAT-001 for 30 minutes
  Interventions: Device: SAT-001
- Modified SAT-001 Treatment Group (Active Comparator): using modified SAT-001, which excludes rest session from SAT-001, for 15 minutes
  Interventions: Device: modified SAT-001

INTERVENTIONS:
Device: SAT-001 — SAT-001 Treatment Group Participants in this group will use the SAT-001 device for 30 minutes. Before and after using the device, choroidal thickness will be measured using Optical Coherence Tomography (OCT) to assess changes in choroidal thickness.
  Arms: SAT-001 Treatment Group
Device: modified SAT-001 — mSAT-001 Treatment Group Participants in this group will use the modified SAT-001 (mSAT-001) device for 15 minutes. Similar to the SAT-001 group, choroidal thickness will be measured using Optical Coherence Tomography (OCT) before and after device usage.
  This protocol will help evaluate the effect of the SAT-001 and modified device on choroidal thickness, with measurements taken before and after each usage.
  Other Names: mSAT-001
  Arms: Modified SAT-001 Treatment Group

SUMMARY:
This clinical trial aims to exploratively compare and evaluate the structural changes in the eye (specifically changes in choroidal thickness) pre- and post-treatment of the investigational medical devices ('SAT-001' and 'modified SAT-001') in pediatric myopia patients, and the differences in their effects on the eye.

DETAILED DESCRIPTION:
Myopia is a rapidly growing global concern, particularly in pediatric populations, with high rates of progression and the potential for serious long-term consequences. The risk of developing high myopia, which can lead to complications such as retinal detachment, cataracts, glaucoma, and optic nerve abnormalities, underscores the importance of effective management strategies for pediatric myopia. While treatments to slow myopia progression have been explored, including pharmacological and non-pharmacological approaches, further investigation is needed into their long-term safety and efficacy.

This multicenter, randomized, open-label, parallel-group, exploratory clinical trial aims to evaluate the impact of SAT-001, a Software as a Medical Device (SaMD), on choroidal thickness in pediatric patients. The study will compare changes in choroidal thickness between two groups: one receiving SAT-001 and the other receiving mSAT-001, a modified version of SAT-001 that excludes the rest period during device use. Participants will be assessed before and after a single application of the device.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 4 to 12
2. Meet the following refractive criteria by cycloplegic refraction

   1. Spherical equivalent refractive error (SER): -0.75 to less than -6.00 D in both eyes
   2. Astigmatism of 2.50 D or less in both eyes
3. Best corrected visual acuity of 0.2 logMAR or better in each eye at the Screening Visit
4. Gestational age of 38 weeks or more at birth, or birth weight of 2,500g or more
5. Transparent ocular media
6. Participants and their legal guardians who agree to participate in the clinical trial and are willing to provide signed informed consent after receiving and understanding the explanation of the trial description (participants under 6 years old may mark their agreement after receiving full information and understanding)

Exclusion Criteria:

1. History of eye diseases such as manifest strabismus, intermittent strabismus, amblyopia, and nystagmus (excluding strabismus that maintains binocular vision)
2. History of ocular surgery such as eyelid surgery, strabismus surgery, intraocular surgery, or refractive correction surgery (excluding simple double eyelid surgery)
3. Ocular abnormalities in cornea, lens, central retina, iris, ciliary body, etc., or presence of malignant tumors in the orbital area
4. History of multifocal lenses (e.g., progressive lenses), corneal refractive therapy lenses (Ortho-K, e.g., Dream lenses), rigid gas permeable (RGP) hard lenses, defocus incorporated multiple segments (DIMS) spectacle lenses (e.g., MyoSmart) within 30 days prior to Visit 2.
5. History of using myopia control agents (e.g., atropine) within 30 days prior to Visit 2
6. Currently participating in another clinical trial or who have participated in another clinical trial within 3 months prior to screening (Visit 1)
7. Inappropriate at the discretion of the investigator due to potential ethical concerns or the possibility of affecting the clinical trial results

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2024-08-19 (Actual); Primary Completion 2024-10-28 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Comparison of change in choroidal thickness from T0 to T1 (without device use) and from T1 to T2 (with device use) in Group 1 | Baseline, 15 minute before device use, 15(mSAT-001 group) or 30(SAT-001 group) minutes after device use
  Choroidal thickness will be measured using Optical Coherence Tomography (OCT) at five points: subfoveal, nasal, and temporal regions. The following comparisons will be made within Group 1:
  Change in Choroidal Thickness from Baseline (T0) to just before SAT-001 application (T1).
  Change in Choroidal Thickness from just before SAT-001 application (T1) to after SAT-001 application (T2).
  These changes will be evaluated and compared within Group 1.
Comparison of change in choroidal thickness change from T0 to T1 (without device use) and from T1 to T2 (with device use) in Group 2 | Baseline, 15 minute before device use, 15(mSAT-001 group) or 30(SAT-001 group) minutes after device use
  Choroidal thickness will be measured using Optical Coherence Tomography (OCT) at five points: subfoveal, nasal, and temporal regions. The following comparisons will be made within Group 2:
  Change in Choroidal Thickness from Baseline (T0) to just before mSAT-001 application (T1).
  Change in Choroidal Thickness from just before mSAT-001 application (T1) to after mSAT-001 application (T2)
Comparison of change in choroidal thickness from T1 to T2 between Group 1 and Group 2 | 15 minute before device use, 15(mSAT-001 group) or 30(SAT-001 group) minutes after device use
  Choroidal thickness will be measured using Optical Coherence Tomography (OCT) at five points: subfoveal, nasal, and temporal regions. The following comparison will be made:
  Comparison of Choroidal Thickness Change from pre- (T1) to post-treatment of application (T2) between Group 1 (SAT-001) and Group 2 (mSAT-001).

CONTACTS AND LOCATIONS:
Overall Officials: Soolienah Rhiu, MD, Principal Investigator — Dongtan Sacred Heart Hospital; So Young Han, MD, Principal Investigator — Kangbuk Samsung Hospital
Locations (2):
- South Korea (2):
  - Hallym University Dongtan Sacred heart Hospital, Hwaseong-si
  - Kangbuk Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No